CLINICAL TRIAL: NCT01222832
Title: Effectiveness of Antibiotic Delivery Via Bio-absorbable Sponge After Functional Endoscopic Sinus Surgery
Brief Title: Effectiveness of Antibiotic Delivery Via Bio-absorbable Sponge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Principal Investigator, Peter Catalano, Chief of Otolaryngology, Steward St. Elizabeth's Medical Center of Boston, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00534
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Paranasal Sinus Disease
MeSH Terms: conditions — Paranasal Sinus Diseases | interventions — Bacitracin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bacitracin (Experimental): Nasopore sponge soaked in Bacitracin, no oral antibiotics
  Interventions: Drug: Bacitracin
- Saline (No Intervention): Nasopore sponge soaked in saline, routine oral antibiotics

INTERVENTIONS:
Drug: Bacitracin — Bacitracin soaked nasopore sponge
  Arms: Bacitracin

SUMMARY:
This study will evaluate the efficacy of a nasopore sponge dressing soaked in Bacitracin VS a sponge soaked in Saline / and the administration of oral antibiotics.

DETAILED DESCRIPTION:
Same as above

ELIGIBILITY:
Inclusion Criteria:

* Patient having primary or revision sinus surgery. Aged 18 years or older.Patients must have middle meatus easily identified. The type of surgery will not be influenced by the participation in this study.

Exclusion Criteria:

* Age less then 18
* Known sensitivity to Bacitracin
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Catalano, MD, Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- St. Elizabeth's Medical Center, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bacitracin: Nasopore sponge soaked in Bacitracin
  Bacitracin: Bacitracin soaked sponge
- Saline: Saline soaked sponge and oral antibiotics
Period: Overall Study
Arm/Group | Bacitracin | Saline
Started | 113 | 113
Completed | 113 | 112
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Saline: Nasopore sponge soaked in saline
- Total: Total of all reporting groups
Arm/Group | Bacitracin | Saline | Total
Number analyzed (Participants) | 113 | 113 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 113 | 113 | 226
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 64 | 64 | 128
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 113 | 113 | 226

OUTCOME MEASURES:

1. Primary Outcome: Rate of Infection
Description: Number of participants without infections on post-op visits 90 days.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Bacitracin: Bacitracin soaked sponge
Arm/Group | Bacitracin | Saline
Number analyzed (Participants) | 113 | 113
Participants | 113 | 113

ADVERSE EVENTS:
Time Frame: 1 year
Description: on case by case bases
Arm/Group | Bacitracin | Saline
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/113
Other Adverse Events (participants affected / at risk) | 0/113 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No